CLINICAL TRIAL: NCT05532891
Title: Bariatric Surgery Provision in Response to the COVID-19 Pandemic: Retrospective Cohort Study of a National Registry
Brief Title: Bariatric Surgery and COVID-19
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Other Study IDs: 010420C19
Record Dates: First submitted 2022-09-07; First posted 2022-09-08 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Bariatric Surgery Candidate
MeSH Terms: conditions — COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-pandemic: Patients that underwent elective bariatric surgery in a control period prior to the pandemic (one year from 1st September 2018).
- Pandemic: Patients that underwent elective bariatric surgery during the pandemic (one year from 1st April 2020)
  Interventions: Other: COVID-19 pandemic

INTERVENTIONS:
Other: COVID-19 pandemic — Pandemic group underwent surgery during the COVID-19 pandemic. Pre-pandemic group underwent surgery prior to the pandemic.
  Groups: Pandemic

SUMMARY:
The National Bariatric Surgical Registry (NBSR) is a prospectively collected database for all patients undergoing elective bariatric surgery in the UK. It was used to identify patients that underwent elective bariatric surgery during the pandemic (one year from 1st April 2020). Characteristics of this group were compared with a pre-pandemic cohort (one year from 1st September 2018).

ELIGIBILITY:
Inclusion Criteria:

All patients listed on National Bariatric Surgical Registry (NBSR) that underwent elective bariatric surgery during the pandemic (one year from 1st April 2020) or prior to the pandemic (one year from 1st September 2018) -

Exclusion Criteria:

- Where a variable was 'not recorded' this point was excluded from analysis. For age, gender, procedure type and provider the records were 100% complete, for BMI at time of surgery there was 5% missing data and for other variables the missing value rate was 2% or lower.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients listed on National Bariatric Surgical Registry (NBSR) that underwent elective bariatric surgery during the pandemic (one year from 1st April 2020) or prior to the pandemic (one year from 1st September 2018)
Sampling Method: Non-Probability Sample
Enrollment: 11545 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery and Cancer, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are restrictions on the availability of data for this study, due to the initial patient consent forms, which only allow the sharing of data for research purposes. Researchers wishing to access an anonymized dataset containing individual participant data can apply to the research data management service at St George's University of London UK (researchdata@sgul.ac.uk), where the data is held in a repository.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-pandemic | Pandemic
Started | 8615 | 2930
Completed | 8615 | 2930
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Detailed analysis was performed for the NHS patients only. This is why the numbers of participants here differs from in overall study group, where both private and NHS records were included.
Groups:
- Pre-pandemic NHS Patients: Patients that underwent elective bariatric surgery in a control period prior to the pandemic (one year from 1st September 2018) in the NHS
- Pandemic NHS Patients: Patients that underwent elective bariatric surgery during the pandemic (one year from 1st April 2020) in the NHS
  COVID-19 pandemic: Pandemic group underwent surgery during the COVID-19 pandemic. Pre-pandemic group underwent surgery prior to the pandemic.
- Total: Total of all reporting groups
Arm/Group | Pre-pandemic NHS Patients | Pandemic NHS Patients | Total
Number analyzed (Participants) | 6384 | 1566 | 7950
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (11.4) | 46.3 (11.6) | 45.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5058 | 1266 | 6324
  Male | 1326 | 300 | 1626
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI at time of surgery kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 45.5 (8.3) | 45.2 (8.3) | 45.4 (8.3)
T2DM on treatment/ pre-T2DM/ no T2DM [Count of Participants; unit: Participants] — Population: A small number of patients did not have this variable recorded
  Participants
    number analyzed (Participants) | 6270 | 1546 | 7816
    T2DM on treatment | 1635 | 397 | 2032
    pre-T2DM | 242 | 72 | 314
    no T2DM | 4393 | 1077 | 5470
Duration of T2DM less than 5 years/ 5-10 years/ more than 10 years; n [Count of Participants; unit: Participants] — Population: This measure only applies to patients with Type 2 Diabetes on treatment (see previous baseline measure) who additionally had data available (some participants had missing data).
  Participants
    number analyzed (Participants) | 1582 | 385 | 1967
    Less than 5 years | 904 | 202 | 1106
    5-10 years | 314 | 83 | 397
    More than 10 years | 364 | 100 | 464
Hypertension [Count of Participants; unit: Participants] — Population: A small number of patients did not have this variable recorded
  Participants
    number analyzed (Participants) | 6272 | 1552 | 7824
    (all) | 2192 | 550 | 2742
Cardiovascular disease [Count of Participants; unit: Participants] — Population: A small number of patients did not have this variable recorded
  Participants
    number analyzed (Participants) | 6261 | 1551 | 7812
    (all) | 307 | 66 | 373
Obstructive sleep apnoea (OSA) [Count of Participants; unit: Participants] — Population: This measure only applies to patients with data for this variable available, a small number of participants did not have this data recorded
  Participants
    number analyzed (Participants) | 6271 | 1553 | 7824
    No indication of OSA | 4511 | 1090 | 5601
    OSA on treatment | 1402 | 400 | 1802
    OSA off treatment | 358 | 63 | 421
Liver disease [Count of Participants; unit: Participants] — Population: A small number of patients did not have this variable recorded
  Participants
    number analyzed (Participants) | 6207 | 1534 | 7741
    (all) | 449 | 110 | 559

OUTCOME MEASURES:

1. Primary Outcome: Revisions
Description: Number of patients undergoing revisional bariatric surgery
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-pandemic | Pandemic
Number analyzed (Participants) | 8615 | 2930
Participants | 746 | 316

2. Primary Outcome: Private
Description: Number of patients undergoing elective bariatric surgery in the private sector
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-pandemic | Pandemic
Number analyzed (Participants) | 8615 | 2930
Participants | 2084 | 1356

3. Secondary Outcome: Completed Laparoscopically
Description: Number of cases completed laparoscopically for patients undergoing elective bariatric surgery in the NHS
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-pandemic NHS Patients | Pandemic NHS Patients
Number analyzed (Participants) | 6280 | 1553
Participants | 6268 | 1552

4. Secondary Outcome: Length of Stay
Description: Length of stay for NHS patients undergoing bariatric surgery in days
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pre-pandemic NHS Patients | Pandemic NHS Patients
Number analyzed (Participants) | 6384 | 1566
days | 2.17 (3.84) | 2.0 (3.43)

5. Secondary Outcome: Surgical Complications
Description: Number of surgical complications in patients undergoing elective bariatric surgery in the NHS
Time Frame: 1 year
Population: refers to NHS patients only, whereas the adverse events tables refer to the population as a whole (NHS and private). Hence the different numbers of participants analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-pandemic NHS Patients | Pandemic NHS Patients
Number analyzed (Participants) | 6384 | 1566
Participants | 126 | 22

6. Secondary Outcome: Presence of Second Consultant
Description: Presence of second consultant in elective bariatric cases undertaken in the NHS
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-pandemic NHS Patients | Pandemic NHS Patients
Number analyzed (Participants) | 6384 | 1566
Participants | 289 | 56

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pre-pandemic | Pandemic
All-Cause Mortality (participants affected / at risk) | 0/8615 | 1/2930
Serious Adverse Events (participants affected / at risk) | 0/8615 | 0/2930
Other Adverse Events (participants affected / at risk) | 151/8615 | 38/2930
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-pandemic (N=8615) | Pandemic (N=2930)
Complication (General disorders) | 151 | 38 — Any complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT05532891/Prot_SAP_000.pdf